CLINICAL TRIAL: NCT03493841
Title: Comparing Gastrointestinal Tolerability and Absorption of Racemic Lipoic Acid and R-lipoic Acid in Progressive Multiple Sclerosis: a Randomized Crossover Trial
Brief Title: Comparing Tolerability and Absorption of Racemic and R-lipoic Acid in Progressive Multiple Sclerosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rebecca Spain (Other)
Responsible Party: Sponsor-Investigator, Rebecca Spain, Principal Investigator, Oregon Health and Science University
Organization: Oregon Health and Science University (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB #17951
Record Dates: First submitted 2018-03-21; First posted 2018-04-11 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Multiple Sclerosis; Progressive Multiple Sclerosis; Secondary Progressive Multiple Sclerosis; Primary Progressive Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Chronic Progressive | interventions — Thioctic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A will receive racemic lipoic acid first and R-lipoic acid second
  Interventions: Drug: Alpha Lipoic Acid
- Group B (Experimental): Group B will receive R- lipoic acid first and racemic lipoic acid second
  Interventions: Drug: Alpha Lipoic Acid

INTERVENTIONS:
Drug: Alpha Lipoic Acid — Lipoic acid is an over the counter supplement. Two different forms, R and racemic are available. R-lipoic acid is the naturally occurring form. Racemic lipoic acid is the most commonly available supplement.
  Other Names: lipoic acid; R-lipoic acid

SUMMARY:
This is a three-week crossover study that will compare how the body absorbs and tolerates two different forms of lipoic acid: R form and racemic form.

DETAILED DESCRIPTION:
This three-week double-blind crossover trial will compare two different forms of lipoic acid (LA). Every participant will take one week of daily oral 600mg R LA, have a one week washout period without LA, and take one week of daily oral 1200mg racemic LA. The order of LA type will be determined by randomization. Blood analyses will be performed to determine which form is better absorbed and a side effects questionnaire will be completed at each visit in order to determine which form is better tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Progressive Multiple Sclerosis
* 18 years of age or older
* Able to give informed consent and adhere to the study activities
* Able to swallow large oral capsules

Exclusion Criteria:

* Clinical Multiple Sclerosis relapse in the prior 1 year
* Oral or IV steroids in the prior 3 months
* Have taken LA in last 30 days
* Clinically significant kidney disease as determined by the PI including, but not limited to, major kidney disease diagnoses, abnormal laboratory values related to renal function, or other related conditions
* Insulin-dependent diabetes
* Other significant ongoing medical illness that may interfere with study procedures
* Taking oral anticoagulants (e.g. Coumadin). Aspirin, clopidogrel, and dipyridamole are acceptable to take
* Pregnant or breast-feeding
* Any condition which would make the patient, in the opinion of the investigator, unsuitable for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-06-08 (Actual); Primary Completion 2019-01-25 (Actual); Study Completion 2019-01-25 (Actual)

PRIMARY OUTCOMES:
Comparison of oral tolerance between R-LA and racemic LA | Obtained at first (Visits 1 and 3) and last doses (visits 2 and 4) of each form of LA. Each visit is approximately a week apart.
  Oral tolerance will be determined by the completion of a modified Monitoring of Side Effects Scale at each study visit. This scale asks the participant to rate the following side effects: abdominal pain, appetite: decreased, appetite: increased, constipation, diarrhea, flatulence, nausea/vomiting, taste abnormality (metallic, etc.), thirst: increased, thirst: decreased, and weight: increased. Each side effect will be rated on severity. 0 - the lowest possible score represents "not present". 4 - the highest possible score represents "severe". The relative change in total tolerance score will be compared between R-LA and racemic LA.
Comparison of serum bioavailability as measured by Area Under the Curve (0-infinity) between R-LA and racemic LA | Obtained at first (Visits 1 and 3) and last doses (visits 2 and 4) of each form of LA. Each visit is approximately a week apart.
  Serum bioavailability, as measured by Area Under the Curve (0-infinity) will be compared between R-LA and racemic LA by obtaining concentration values at times 0, 60, 90, 120, 180, and 240 minutes after ingestion of LA dose on the first (visits 1 and 3) and last doses (visits 2 and 4) of each LA form.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Spain, MD, MSPH, Principal Investigator — Oregon Health and Science University; Michelle Cameron, MD, PT, MCR, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States